CLINICAL TRIAL: NCT05829629
Title: Randomised, Double-blind, Placebo-controlled Phase 1 Dose-escalation Study of FluBHPVE6E7 in HPV16-infected Women with NILM, ASC-US, LSIL or Low-grade CIN
Brief Title: Phase 1 Dose-escalation Study of FluBHPVE6E7 in HPV16-infected Women
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BlueSky Immunotherapies GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BS-02
Record Dates: First submitted 2023-04-11; First posted 2023-04-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: HPV Infection; HPV-Related Cervical Carcinoma
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FluBHPVE6E7 (Experimental): intracervical and intramuscular 0.5 ml per dose 3 doses (12 weeks)
  Interventions: Biological: FluBHPVE6E7
- Placebo (Placebo Comparator): intracervical and intramuscular 0.5 ml per dose 3 doses (12 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: FluBHPVE6E7 — Intracervical administration for first dose followed by intramuscular administration for subsequent doses at recommended dose level and determined schedule
  Arms: FluBHPVE6E7
Drug: Placebo — Intracervical administration for first dose followed by intramuscular administration for subsequent doses at determined schedule
  Arms: Placebo

SUMMARY:
BS-02 is a randomised, double-blind, placebo-controlled, phase 1 dose escalation study to assess the safety, tolerability and immunogenicity of FluBHPVE6E7, in women infected with HPV-16. with cervical cytological evaluation negative for intraepithelial lesion or malignancy (NILM), atypical squamous cells of undetermined significance (ASC-US), low grade squamous intraepithelial lesion (LSIL), or low-grade cervical intraepithelial neoplasia (CIN1).

DETAILED DESCRIPTION:
FluBHPVE6E7 is an influenza virus vector that was modified on several levels to be used as an immunotherapeutic agent against human papillomavirus (HPV) infections, and precancers and cancers induced by HPV.

Study BS-02 investigates the safety, tolerability and immunogenicity of FluBHPVE6E7 in HPV-16 infected women.

FluBHPVE6E7 is administered three times at two dose levels. The first dose is administered into the cervix, subsequent doses are administered intramuscularly.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18-49 years of age with HPV16 infection and cervical cytological evaluation negative for intraepithelial lesion or malignancy (NILM), atypical squamous cells of undetermined significance (ASC-US), low grade squamous intraepithelial lesion (LSIL), or low-grade cervical intraepithelial neoplasia (CIN1)
* HPV16 infection has been confirmed at least twice by a validated HPV test separated by at least 3 months
* Satisfactory colposcopy
* No clinically significant out of range haematological, renal or hepatic laboratory tests
* Normal screening ECG or screening ECG with no clinically significant findings, as judged by the investigator
* Negative serum pregnancy test at screening
* Agree to use a reliable form of contraception during the whole study period.
* Provides written informed consent

Exclusion Criteria:

* Any vaccination within 6 weeks of day 0
* Active significant viral infections including influenza, CMV, and EBV within 30 days of receiving study treatment
* Co-infection with hepatitis B, hepatitis C, or HIV or having other immune deficient states
* Current Bacterial Vaginosis (BV) infection
* Current high-grade cervical intraepithelial neoplasia (CIN2/3)
* Prior history of or current malignancy, vulvar intraepithelial neoplasia (VIN), vaginal intraepithelial neoplasia (VAIN), atypical glandular cells (AGC), adenocarcinoma in situ (AIS) or any suspicion of either micro-invasive or invasive disease
* Pregnancy, breastfeeding
* Influenza-like illness (ILI) within 3 months of day 0
* Known hypersensitivity to oseltamivir or any of its components
* Any anatomical condition of the cervix, including that resulting from previous cervical surgery, congenital malformation or other condition, that would interfere with a complete evaluation of the cervix
* Current pelvic inflammatory disease, cervicitis, or other gynaecological infection as per colposcopy and clinical examination
* Serious, concomitant disorder, including active systemic infection requiring treatment
* Presence of acute or chronic bleeding or clotting disorder, or use of blood thinners within 2 weeks of day 0
* A proven or suspected autoimmune disease
* Immunosuppression including any concurrent condition requiring the continued use of systemic or topical steroids, or the use of immunosuppressive agents, disease modifying doses of anti-rheumatic drugs, and biologic disease modifying drugs. Any immunosuppressive agents containing corticosteroids or monoclonal antibodies specific for the treatment of obstructive airway, ear or vestibular diseases are permissible.
* Acute or history of Herpes genitalis
* Prior major surgery within 4 weeks of day 0
* Administration of any blood product within 3 months of enrolment
* Any current significant cardiac, hepatic or renal disease or history of clinically significant, medically unstable disease
* Any current or history of neurological disease including history of seizures
* Participation in another experimental protocol/use of investigational drug during the prior two months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants are assigned females at birth.
Enrollment: 20 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) | 7 days
  The severity of the adverse event is assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

SECONDARY OUTCOMES:
Induction of HPV-specific T-cell response following FluBHPVE6E7 administration | 16 weeks
  To evaluate the induction of HPV16 E6- and E7-specific T-cells (%) by IFN-gamma ELISPOT analysis.
Hemagglutination Inhibition (HAI) Geometric Mean Titers (GMTs) following FluBHPVE6E7 administration | 16 weeks
  To evaluate the induction of systemic vector-specific antibodies by HAI assay.
Local HPV clearance | 16 weeks
  To evaluate the status of HPV-16 infection by HPV test (yes or no).
Cervical cytology | 16 weeks
  To evaluate changes in cervical cytology by Pap smear. Results are reported as Pap results according to the Bethesda System.
Biodistribution: Detection of FluBHPVE6E7 in blood samples | 16 weeks
  To evaluate the presence of FluBHPVE6E7 by quantification of FluBHPVE6E7 genome copies in blood samples by RT-qPCR (copies per ml blood).
Biodistribution: Detection of FluBHPVE6E7 in saliva | 16 weeks
  To evaluate the presence of FluBHPVE6E7 by qualitative real-time PCR assay specific for influenza B virus (positive or negative).
Viral shedding: Detection of FluBHPVE6E7 in vaginal secretion samples | 16 weeks
  To evaluate the presence of FluBHPVE6E7 by quantification of FluBHPVE6E7 genome copies in vaginal secretion samples by RT-qPCR (copies per sample).
Number of participants with adverse events (type, frequency, severity). | 16 weeks
  To assess the safety and tolerability of FluBHPVE6E7 by monitoring the type, frequency, and severity of AEs.

CONTACTS AND LOCATIONS:
Locations (1):
- Univerzitná nemocnica Bratislava, Bratislava, Slovakia